CLINICAL TRIAL: NCT02193854
Title: Teledermatology Solution Through Mobile Phone in Rural Mongolia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: Health Science University of Mongolia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: TaipeiMU
Record Dates: First submitted 2014-06-09; First posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Social Distance
Keywords: Telemedicine; Mobile phone; Rural physicians; Mongolia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mobile phone (Experimental): General practitioners (GPs) received TD consultation through Sana system.
  Mobile phones with Sana system installed were provided to 10 rural GPs from three different districts of Mongolia.
  Interventions: Device: Mobile Phone

INTERVENTIONS:
Device: Mobile Phone — Investigators used Sana system, that is a mobile phone-based, open source software platform for telemedicine services. The Android-based system supports multimedia, location-based data, and text. In the village health clinic, a healthcare worker will interact with a patient and collects data through a step-by-step clinical questionnaire on a smart mobile phone. As patients' data is uploaded to an open source electronic medical record system (OpenMRS) with a diagnosis-specific information and images. The consultant can access the clinical information about the patient and make appropriate diagnoses and treatment recommendations from the secondary hospital.

SUMMARY:
Objective This study is aimed to estimate the distance, time and the cost of travel saved by patients who are seeking tele-dermatology (TD) service though smart mobile phones in the resource poor settings at the rural clinics of Mongolia.

Methods A cluster-randomised trial was conducted for six months at the 20 rural health clinics selected from three districts in Mongolia. With a computer-generated sequence, health clinics were randomly allocated either to the intervention group, in which all general practitioners (GPs) received TD consultation through Sana system, or the control group, in which GPs referred patients to the dermatologist at district hospital whenever needed. The primary outcome was to estimate the distance traveled, times spend and the cost of travel required in receiving dermal care for patients in rural Mongolia. Analysis was done to estimate the difference between the aforementioned parameters among intervention and control groups.

DETAILED DESCRIPTION:
The investigators used Sana system, that is a mobile phone-based, open source software platform for telemedicine services. The Android-based system supports multimedia, location-based data, and text. In the village health clinic, a healthcare worker will interact with a patient and collects data through a step-by-step clinical questionnaire on a smart mobile phone. As patients' data is uploaded to an open source electronic medical record system (OpenMRS) with a diagnosis-specific information and images. The consultant can access the clinical information about the patient and make appropriate diagnoses and treatment recommendations from the secondary hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-98 years visiting with dermal problem.

Exclusion Criteria:

* Patients who do not need dermal care.
* Patients who are already under treatment for dermal problem.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2013-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Comparison between the number of referrals in the control and intervention groups | up to 5 months
  Outcome measures are the number of referrals done in the control and in the intervention groups. We compared the difference in the number of referrals with Sana system and without.

SECONDARY OUTCOMES:
Satisfaction by physicians and patients by questionnaire | up to 5 months
  Both physicians and patients who were in the intervention group were satisfied by the Sana system.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chuan Li, MD., PhD., Principal Investigator — Taipei Medical University
Locations (1):
- Shabbir Syed Abdul, Taipei, Taipei, Taiwan

REFERENCES:
- See also: International Center for Health Information Technologies — http://ichit.tmu.edu.tw